CLINICAL TRIAL: NCT00819221
Title: A Phase I, Open Label, Multicenter Study to Assess the Safety, Tolerability and Pharmacology of AZD2281 in Combination With Liposomal Doxorubicin (Caelyx®) in Patients With Advanced Solid Tumors
Brief Title: AZD2281 in Combination With Liposomal Doxorubicin in Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0810L00001; Eudract No. 2008-007680-17
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumors
Keywords: advanced tumors; solid tumors; dose escalation; combination; AZD2281; liposomal doxorubicin; pharmacology; phase I; multicenter
MeSH Terms: interventions — olaparib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD2281; Drug: liposomal doxorubicin

INTERVENTIONS:
Drug: AZD2281 — capsules, oral, bd, 2 months
  Other Names: Olaparib
Drug: liposomal doxorubicin — once every 4 weeks at 40mg/m2

SUMMARY:
The study will be an open label, multicenter, dose finding study. Depending on the tolerated dose up to 7 dose levels will be explored in this study, approximately 33 patients (21-54 depending on number of cohorts) may be enrolled into this study. Three patients will be initially dosed in each cohort. The primary objective of this study is to determine the recommended dose (RD) of twice daily oral doses of AZD2281 either as intermittent therapy for 7 days out of a 28-day schedule or given continuously, administered in combination with liposomal doxorubicin to patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic cancer, not amenable to surgery or radiation therapy with curative intent
* Measurable or evaluable disease
* ECOG Performance status 0 - 2
* Estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* More than 3 prior lines of chemotherapy for advanced disease
* Less than 28 days from active treatment (ie, any treatment used to treat the disease) or high dose radiotherapy (patients may continue concomitant use of stable dose of bisphosphonates if used at least 28 days prior to commencing study treatment and pat
* Prior treatment with >300mg/m2 cumulative dose of doxorubicin equivalent
* Resistance to anthracyclines defined as progressive disease during anthracycline treatment or within 6 months after the last anthracycline administration.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-01-05 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
recommended dose | 2 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 visits within 1 month
safety/tolerability/toxicity | 2 months
DNA repair mechanism | once

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca
Locations (3):
- Research Site, Milan, Italy
- Switzerland (2):
  - Research Site, Bellinzona
  - Research Site, Chur

REFERENCES:
- [Derived] Del Conte G, Sessa C, von Moos R, Vigano L, Digena T, Locatelli A, Gallerani E, Fasolo A, Tessari A, Cathomas R, Gianni L. Phase I study of olaparib in combination with liposomal doxorubicin in patients with advanced solid tumours. Br J Cancer. 2014 Aug 12;111(4):651-9. doi: 10.1038/bjc.2014.345. Epub 2014 Jul 15. PMID 25025963
- See also: Study protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1679&filename=Swiss_Study_Protocol_excl_personal_info_SECURE.pdf
- See also: D0810L00001_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1679&filename=D0810L00001.pdf